CLINICAL TRIAL: NCT03794154
Title: A PHASE IV, SINGLE-DOSE, OPEN-LABEL, RANDOMIZED, 2-WAY CROSSOVER STUDY TO DETERMINE THE BIOEQUIVALENCE OF DULOXETINE HYDROCHLORIDE HARD GELATINOUS CAPSULE WITH DELAYED RELEASE MICROGRANULES (60 MG; PFIZER S.R.L - ARGENTINA.) COMPARED TO CYMBALTA (REGISTERED) MICROGRANULES (60 MG; ELI LILLY DO BRASIL LTDA) IN HEALTHY MALE RESEARCH SUBJECTS UNDER FED CONDITIONS
Brief Title: A Study Of Duloxetine Hydrochloride Hard Gelatinous Capsule Compared To Cymbalta Under Fed Conditions
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study has been cancelled prior to FSFV due to business reasons
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B2781005
Record Dates: First submitted 2018-12-20; First posted 2019-01-04 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — Duloxetine Hydrochloride; Drug Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine hydrochloride (Experimental): Duloxetine hydrochloride hard gelatinous capsule 60 mg by mouth on Day 1 of period 1 or 2
  Interventions: Drug: Duloxetine hydrochloride capsule
- Cymbalta (Active Comparator): Duloxetine hydrochloride hard gelatinous capsule 60 mg as Cymbalta by mouth on Day 1 of period 1 or 2
  Interventions: Drug: Cymbalta capsule

INTERVENTIONS:
Drug: Cymbalta capsule — Active Comparator: Cymbalta®- hard gelatinous capsule with delayed release microgranules ( Eli Lilly do Brasil Ltda) equivalent to 60 mg of duloxetine.
  Other Names: Reference drug
  Arms: Cymbalta
Drug: Duloxetine hydrochloride capsule — Experimental Drug: Duloxetine hydrochloride - hard gelatinous capsule with delayed release microgranules (Pfizer S.R.L - Argentina.) equivalent to 60 mg of duloxetine.
  Other Names: Test drug
  Arms: Duloxetine hydrochloride

SUMMARY:
In Brazil, duloxetine is currently available as hard gelatinous capsule with delayed release microgranules for oral administration containing enteric-coated pellets of 33.7, or 67.3 mg of duloxetine hydrochloride equivalent to 30 mg or 60 mg of duloxetine (Cymbalta®), respectively.

The Sponsor has developed a hard gelatinous capsule with delayed release microgranules formulation containing enteric-coated pellets of 33.7, or 67.3 mg of duloxetine hydrochloride equivalent to 30, or 60 mg of duloxetine, respectively.

The purpose of this study is to verify through a single dose study, if the test formulation of duloxetine is bioequivalent to the reference formulation (Cymbalta®) when administered with the same dosage and under fed conditions in healthy male research subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male research subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive.
* Body mass index (BMI) of 18.5 kg/m2 to 24.9 kg/m2, and a total body weight >50 kg (>110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the research subject has been informed of all pertinent aspects of the study.
* Research subjects that never smoked.
* Research subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Clinically significant infections within the past 3 months, evidence of any infection within the past 7 days, history of disseminated herpes simplex infection or recurrent (>1 episode) or disseminated herpes zoster.
* Vaccination with live or attenuated vaccines within 6 weeks prior to dosing.
* A history of suicidal thoughts, behavior or suicide attempts.
* History of narrow angle glaucoma.
* Any condition possibly affecting drug absorption (eg, gastrectomy, colon resection, etc.).
* History of or current positive results for any of the following serological tests: hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), anti hepatitis C core antibody (HCV Ab), or human immunodeficiency virus (HIV) 1 and 2.
* Malignancy or a history of malignancy.
* A positive urine drug test.
* A positive alcohol screen.
* History of regular alcohol consumption exceeding 21 drinks/week for male research subjects [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months before screening.
* Use of tobacco or all nicotine containing products.
* Treatment with an investigational drug within 6 months or 5 half lives preceding the first dose of investigational product (whichever is longer).
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Use of prescription or nonprescription drugs and dietary supplements within 14 days or 5 half lives (whichever is longer) prior to the first dose of investigational product.
* Consumption of grapefruit or grapefruit related citrus fruits (eg, Seville oranges, pomelos) or juices within 7 days prior to dosing.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 3 months prior to screening until collection of the final PK blood sample (Period 2, Day 4).
* History of sensitivity to heparin or heparin induced thrombocytopenia.
* History of hypersensitivity to duloxetine or any of the components in the formulation of the study products.
* Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
* Use of any medicinal product that is an inductor or strong inhibitor of CYP450 1A2 or 2D6 (eg, rifampicin, omeprazole, fluvoxamine, ciprofloxacin, fluoxetine, paroxetine, etc) within two weeks before administration of the investigational product and at any time during the study.
* Use of any medicinal product that inhibits monoamine oxidase A or B (eg, phenelzine, isocarboxacid, linezolid) within two weeks before administration of the investigational product and at any time during the study till at least 5 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2020-06-05 (Estimated); Study Completion 2020-06-05 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve | Upto 72 hours post dose
  Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast)
Maximum plasma concentration (Cmax) | Upto 72 hours post dose

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero extrapolated to infinite time | Upto 72 hours post dose
Time to first occurrence of Cmax (Tmax) | Upto 72 hours post dose
Terminal phase rate constant (kel) | Upto 72 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2781005&StudyName=A+Phase+Iv%2C+Single-dose%2C+Open-label%2C+Randomized%2C+2-way+Crossover+Study+To+Determine+The+Bioequivalence+Of+Duloxetine+Hydrochloride+Hard+Gelatinous+Capsule+With+Delayed+Release+Microgranules+%2860+Mg%3B+Pfizer+S.r.l+-+Argentina.%29+Compared+To+Cymbalta+%28registered%29%EF%83%92microgranules+%2860+Mg%3B+Eli+Lilly+Do+Brasil+Ltda%29+In+Healthy+Male+Research+Subjects+Under+Fed+Conditions
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2781005&StudyName=A+Phase+Iv%2C+Single-dose%2C+Open-label%2C+Randomized%2C+2-way+Crossover+Study+To+Determine+The+Bioequivalence+Of+Duloxetine+Hydrochloride+Hard+Gelatinous+Capsule+With+Delayed+Release+Microgranules+%2860+Mg%3B+Pfizer+S.r.l+-+Argentina.%29+Compared+To+Cymbalta+%28registered%29+Microgranules+%2860+Mg%3B+Eli+Lilly+Do+Brasil+Ltda%29+In+Healthy+Male+Research+Subjects+Under+Fed+Conditions
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2781005&StudyName=A+PHASE+IV%2C+SINGLE-DOSE%2C+OPEN-LABEL%2C+RANDOMIZED%2C+2-WAY%0ACROSSOVER+STUDY+TO+DETERMINE+THE+BIOEQUIVALENCE+OF%0ADULOXETINE+HYDROCHLORIDE+HARD+GELATINOUS+CAPSULE+WITH%0ADELAYED+RELEASE+MICROGRANULES+%2860+MG%3B+PFIZER+S.R.L+-+ARGENTINA.%29+COMPARED+TO+CYMBALTA+%28REGISTERED%29+MICROGRANULES+%2860+MG%3B+ELI+LILLY+DO+BRASIL+LTDA%29+IN+HEALTHY+MALE+RESEARCH+SUBJECTS+UNDER+FED+CONDITIONS